CLINICAL TRIAL: NCT06725953
Title: Cerebrovascular, Cognitive, Pro-Inflammatory, and Cardiometabolic Outcomes in Cancer Survivors With and Without Type II Diabetes Reporting Chemo-Brain: Baseline Differences and Impact of Activity
Brief Title: Remote Physical Activity Programming to Improve Outcomes in Cancer Survivors With and Without Type 2 Diabetes
Acronym: CICI-PA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17332; HR23-061-2 (Other Grant/Funding Number: Harold Hamm Diabetes Center-Stephenson Cancer Center Team Science Grant)
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Cancer Survivorship; Chemotherapy Side Effects
Keywords: Aerobic Physical Activity; Resistance Training; Wearable Devices; Smartphone Applications; Cancer Survivors; Chemo-Brain; Health Outcomes

STUDY DESIGN:
Intervention Model Description: Social Cognitive Theory-based, Technology-delivered Physical Activity Program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Social Cognitive Theory-based, Technology-delivered Physical Activity Program (Experimental): Participants will engage in a 12-week program of aerobic and muscle-strengthening physical activity. This program will be delivered remotely via two smartphone applications--one for providing health education, goal setting, and journaling features and the other for delivery of the physical activity program in a highly-personalized and HIPAA-compliant manner. Participants will receive a Fitbit to track their activity and resistance bands to use during their resistance training physical activity. All program components will be based in the Social Cognitive Theory and will target improving participants' physiological and psychological health outcomes.
  Interventions: Behavioral: Social Cognitive Theory-based, Technology-delivered Physical Activity Program

INTERVENTIONS:
Behavioral: Social Cognitive Theory-based, Technology-delivered Physical Activity Program — Participants will engage in a 12-week program of aerobic and muscle-strengthening physical activity. This program will be delivered remotely via two smartphone applications--one for providing health education, goal setting, and journaling features and the other for delivery of the physical activity program in a highly-personalized and HIPAA-compliant manner. Participants will receive a Fitbit to track their activity and resistance bands to use during their resistance training physical activity. All program components will be based in the Social Cognitive Theory and will target improving participants' physiological and psychological health outcomes.

SUMMARY:
The growing U.S. cancer survivor population is projected to hit 26M by 2040. Chemotherapy represents an effective cancer treatment but can diminish cancer survivors' quality of life-particularly cognitive function-through select pathophysiological processes. Research on chemotherapy-induced cognitive impairment (hereafter, 'chemo-brain') is therefore critical. Chemotherapy disrupts immune system function and antioxidant regulation, causing inflammatory molecule release and damaging the brain's blood vessels. The brain's vascular function and, possibly, its neurons, are subsequently impaired-likely contributing to chemo-brain. Type 2 diabetes (T2D), a common cancer survivor comorbidity, shares underlying pathophysiology with chemo-brain. T2D-related insulin resistance can precipitate repeated high blood sugar episodes which increase inflammatory molecule release. In individuals with T2D without cancer, negative relationships are observed between inflammatory molecule concentrations and the brain's vascular and/or cognitive function. Cancer survivors with T2D might thus have higher chemo-brain risk than those without T2D. Yet, more research must compare how the brain's vascular function, as well as cognitive, inflammatory, and cardiometabolic indices, differ between these groups. Physical activity (PA) counteracts chemo-brain's and T2D's pathophysiology, with higher PA/fitness resulting in better vascular function of the brain, lower inflammatory molecule concentrations, and improved insulin sensitivity. We are therefore conducting a 30-participant quasi-experimental pilot study in cancer survivors with (cases) and without (controls) T2D. We will first investigate between-group differences in the brain's vascular function as well as cognitive, inflammatory, cardiometabolic, and epigenetic outcomes. We will then examine between-group changes in these outcomes and select psychosocial metrics during a 12-week technology-based PA program-potentially further elucidating involved mechanisms.

DETAILED DESCRIPTION:
While incident cancer cases of any site remain stable, 5-year cancer survival rates have increased. In January 2022, >18M individuals in the U.S. were CS-reflecting those diagnosed with cancer until death-with a projected increase to 26M by 2040. Although modern cancer treatments are effective, these treatments can worsen CS HRQoL. Several cancer treatments-most notably, chemotherapy-are associated with cognitive difficulties. While chemotherapy effectively treats many malignancies, it also negatively impacts vascular endothelial cells-leading to pathophysiological processes contributing to CS's oft-reported 'chemo-brain' during/after treatment. As CS populations grow, CICI mitigation research is crucial to improve HRQoL.

CICI likely occurs for several reasons. Chemotherapy can induce immune and antioxidant dysregulation. This dysregulation can lead to peripheral pro-inflammatory cytokines being released which damage and cross the blood-brain barrier-contributing to central pro-inflammatory cytokine release and causing neuroinflammation-related impairments in neurogenesis and the myelination process. Endothelial dysfunction and cerebral autoregulation failure can also result from this damage. Reviews suggest these mechanisms alter cerebrovascular function more broadly by impairing cerebral perfusion, glucose metabolism, and angiogenesis; thus contributing to CICI. T2D is both a risk factor for developing several common cancers and, given its prevalence, a common CS comorbidity heightening cancer recurrence risk. Several pathophysiological mechanisms underlying CICI are observed with T2D. Insulin resistance can result in repeated hyperglycemic episodes and subsequent pro-inflammatory cytokine elevation-possibly explaining why insulin resistance is correlated with diminished cerebrovascular and cognitive function in individuals with T2D. This might also explain why, in newly diagnosed CS with pro-inflammatory comorbidities (e.g., T2D), higher pro-inflammatory cytokines and poorer cognitive function have been observed relative to CS without comorbidities-even prior to chemotherapy. CICI mitigation research should thus focus on CS most vulnerable to CICI (e.g., CS with T2D).

Aerobic PA and resistance training (RT) have robust health benefits counteracting much of the pathophysiology underlying CICI and T2D. Reviews suggest better cerebrovascular function in those who are more active and/or fitter relative to those less active and/or fit, with greater fitness positively associated with cognitive function in other at-risk populations. In those with T2D, research has shown that PA is impactful at lowering pro-inflammatory cytokines and improving insulin sensitivity. Yet, research is needed on how increasing PA in CS with T2D reporting CICI improves cerebrovascular and cognitive health through improved fitness.

We are thus conducting a 30-participant quasi-experimental pilot study in CS+T2D (n=15; cases) and CS (n=15; controls)-all self-reporting CICI. We will first investigate cerebrovascular, cognitive, pro-inflammatory, cardiometabolic, and epigenetic (exploratory) differences between CS+T2D and CS given that no known investigations have directly compared these outcomes concurrently between these groups (Aim 1). We will then examine differential between-group changes in these outcomes and select psychosocial metrics during a 12-week technology-delivered PA program grounded in the Social Cognitive Theory-crucial to further investigate how to intervene and reverse the underlying pathophysiology (Aims 2 and 3). This collaboration between clinical scientists and translational researchers is critical to conducting this comprehensive project given our diverse skillsets and preliminary studies. This collaboration will serve our larger goal of acquiring extramural funding to investigate in even greater detail the most clinically-relevant pathophysiological mechanisms observed during this project. Our Aims/Hypotheses are (main outcomes underlined):

Aim 1: Characterize cerebrovascular function, cognitive function, pro-inflammatory cytokines, and cardiometabolic outcome differences between CS+T2D and CS. Our Hypotheses 1 are that CS+T2D will have a: poorer measures of middle cerebral artery velocity and cerebrovascular conductance, reactivity, and resistance. b: lower executive function scores. c: higher c-reactive protein, interleukin-6, and monocyte chemoattractant protein 1 concentrations. and d: higher blood pressure and insulin resistance measures.

Aim 2: Examine pre- to post-PA program differences for changes in A1's cerebrovascular function, cognitive function, pro-inflammatory cytokines, and cardiometabolic outcomes between CS+T2D and CS. Hypothesis 2: We will observe greater pre- to post-PA program improvements in these outcomes for CS+T2D relative to CS.

Aim 3: Assess pre- to post-PA program differences for changes in Social Cognitive Theory (SCT)-based constructs, select psychosocial outcomes, HRQoL, and PA between CS+T2D and CS. Our Hypotheses 3 are that CS+T2D and CS will have similar improvements in a: SCT-based, PA-related self-efficacy, outcome expectancy, enjoyment, social support, and barriers and b: stress, anxiety, mood, and depressive symptoms but that CS+T2D will have greater improvements than CS in c: HRQoL due to greater improvements in physical functioning and pain intensity/interference and d: overall PA participation due to greater increases in light and moderate PA.

Exploratory Aim: Characterize epigenetic markers of biologically-relevant pathways related to neurocognition, energy metabolism, and/or T2D among CS+T2D and CS as well as whether changes are observed in these markers pre- to post-PA program. Exploratory Hypothesis: Distinct epigenetic profiles will be evident between CS+T2D and CS, with both groups experiencing pre- to post-PA program changes in these profiles.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old
2. ability to speak/read English
3. ability to provide informed consent
4. underwent treatment within the last three years for a non-central nervous system-related cancer with said treatment having included chemotherapy
5. self-reported cognitive difficulties following cancer treatment
6. For CS+T2D: current T2D diagnosis as classified by a fasted blood glucose of ≥126 mg/dL, 2-hour oral glucose tolerance test of ≥200 mg/dL, HbA1c level of ≥6.5%, or use of medications to treat hyperglycemia (e.g., Metformin) or For CS: no current T2D diagnosis as classified by a fasted blood glucose <100 mg/dL, 2-hour oral glucose tolerance test <140 mg/dL, or HbA1c level of <5.7%. Presence/absence of T2D to be confirmed preferentially via physician's documentation
7. own smartphone and/or computer with internet access
8. willing to participate in the 12-week remotely-delivered PA program

Exclusion Criteria:

1. reporting a Physical Activity Readiness Questionnaire (2017 PAR-Q) score that indicates PA may potentially be unsafe, unless the participant produces a signed doctor's note. We will define 2017 PAR-Q+ scores as indicating that PA may potentially be unsafe as responding "Yes" to any of the follow-up questions except [1] if the individual indicates that they have high blood pressure but subsequent responses indicate that they do not have problems keeping it under control and that their resting blood pressure is less than 160/90 mmHg, and [2] if the individual indicates that they have a metabolic condition but subsequent responses indicate that they do not have problems controlling their blood sugar levels, do not any experience signs or symptoms of hypoglycemia, and do not have any signs of symptoms of listed diabetes complications)
2. engaging in ≥75 min/week of vigorous-intensity PA, ≥150 min/week of moderate-intensity PA, or an equivalent combination of both over the last 3 months
3. currently a prisoner, pregnant, or planning to become pregnant during study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Middle Cerebral Artery Velocity | Baseline and After Study Week 12
  We will complete transcranial doppler assessments to measure middle cerebral artery velocity at rest and during exercise.
Cerebrovascular Resistance | Baseline and After Study Week 12
  We will complete transcranial doppler assessments to measure cerebrovascular resistance at rest and during exercise.
Cerebrovascular Conductance | Baseline and After Study Week 12
  We will complete transcranial doppler assessments to measure cerebrovascular conductance at rest and during exercise.
Cerebrovascular Pulsatility | Baseline and After Study Week 12
  We will complete transcranial doppler assessments to measure cerebrovascular pulsatility at rest and during exercise.
Dynamic Cerebral Autoregulation | Baseline and After Study Week 12
  We will assess dynamic cerebral autoregulation using the Thigh Cuff Release Challenge technique. Large bilateral blood pressure thigh cuffs are rapidly inflated (rapid cuff inflation/deflation system) to occlude the lower limbs. Blood flow will be monitored in the dorsalis pedis artery, and the initial thigh cuff pressure will start at 20 mmHg above systolic blood pressure. If blood flow is still detected, thigh cuff pressure will increase gradually until occlusion is confirmed. The occlusion will be held for 2 min. After 2 min of occlusion, the cuff pressure is rapidly deflated.
Cognitive Function | Baseline and After Study Week 12
  We will assess cognitive function using the NIH Toolbox-a platform for low-burden, standardized delivery of cognitive function testing. We will employ the NIH Toolbox Cognitive Battery to obtain a Fluid Composite score from all or some of the following five tests: 1) Dimensional Change Card Sort [executive function]; 2) Pattern Comparison Processing Speed; 3) List Sorting Working Memory; 4) Flanker Inhibitory Control and Attention; and/or 5) Picture Sequencing Memory. We will score tests per established standards used in other studies employing NIH Toolbox.

SECONDARY OUTCOMES:
Blood Pressure | Baseline and After Study Week 12
  After five minutes of quiet seated rest, we will take blood pressure measurements in triplicate using an blood pressure cuff around the left arm, with readings separated by 30-second breaks and the lowest two blood pressure readings averaged.
Body Mass Index | Baseline and After Study Week 12
  Body weight and height will be measured using a digital weight scale and stadiometer, respectively, while participants wear disposable hospital gowns. These measurements will be used to calculate body mass index.
Waist-to-Hip Ratio | Baseline and After Study Week 12
  Waist and hip circumference will be assessed per established standards. These measurements will be used to calculate waist-to-hip ratio.
Cholesterol Levels | Baseline and After Study Week 12
  We will complete blood draws to discern cholesterol levels, including high- and low-density lipoprotein and total cholesterol. Reporting these cholesterols simultaneously is commonplace.
Fasting Blood Glucose | Baseline and After Study Week 12
  We will complete blood draws to discern fasting blood glucose levels.
Interleukin-6 | Baseline and After Study Week 12
  We will complete blood draws to discern interleukin-6 levels--a pro-inflammatory marker implicated in chemotherapy-induced cognitive impairment.
Monocyte Chemoattractant Protein 1 | Baseline and After Study Week 12
  We will complete blood draws to discern monocyte chemoattractant protein 1 levels--a pro-inflammatory marker implicated in chemotherapy-induced cognitive impairment.

OTHER OUTCOMES:
Self-Efficacy for Physical Activity | Baseline, After Study Week 6, and After Study Week 12
  Self-efficacy will be assessed using a 9-item measure from Rodgers et al. Participants will note their confidence during different physical activity-related situations ('0%: Not confident at all' to '100%: Extremely confident'; 10% increments).
Social Support for Physical Activity | Baseline, After Study Week 6, and After Study Week 12
  Social support will be evaluated using the Social Support and Exercise Survey, with participants reporting frequency of physical activity support over the last three months from family and, separately, friends ('1: None' to '5: Very often').
Enjoyment of Physical Activity | Baseline, After Study Week 6, and After Study Week 12
  Physical activity-related enjoyment will be measured via the 18-item Physical Activity Enjoyment Scale, with feelings related to physical activity-related statements/situations reported on a 7-point scale (varied response options).
Barriers to Physical Activity | Baseline, After Study Week 6, and After Study Week 12
  We will use a 14-item scale to assess agreement between hypothetical physical activity barriers and participants' perceived barriers ('1: Strongly disagree' to '4: Strongly agree').
Outcome Expectations of Physical Activity | Baseline, After Study Week 6, and After Study Week 12
  The 13-item Outcome Expectations for Exercise Scale-2 will assess agreement with listed positive and negative benefits of physical activity ('1: strongly agree' to '5: strongly disagree').
Perceived Stress | Baseline, After Study Week 6, and After Study Week 12
  We will assess chronic stress with the 10-item Cohen's Perceived Stress Scale. Participants will report stress frequency over the last month ('0: Never' to '4: Very often').
Perceived Anxiety | Baseline, After Study Week 6, and After Study Week 12
  We will measure chronic anxiety with the State-Trait Anxiety Inventory which includes 20 items each on state and trait anxiety ('1: Almost never' to '4: Almost always').
Mood | Baseline, After Study Week 6, and After Study Week 12
  Chronic mood will be assessed by the Positive and Negative Affect Scale. This scale has 10 items each for positive and negative affect ('1: Very slightly or not at all' to '5: Extremely').
Depressive Symptoms | Baseline, After Study Week 6, and After Study Week 12
  Chronic depressive symptoms will be assessed by the 9-item Patient Health Questionnaire-9 ('0: Not at all' to '3: Nearly every day').
Health-related Quality of Life | Baseline, After Study Week 6, and After Study Week 12
  The following components of physical and psychological health will be assessed using the Patient-Reported Outcomes Measurement Information System--allowing us to ascertain a health-related quality of life index measurement: physical functioning, fatigue, anxiety, depression, pain interference, pain intensity, sleep impairment, and sleep disturbance. Measurements are on a 5-point scale, with 5 being worst on all components aside from physical function where higher scores are better.
Overall Physical Activity | Baseline, After Study Week 6, and After Study Week 12
  We will assess physical activity using ActiGraph wGT3X-BT accelerometers-valid for free-living physical activity assessments. Participants will wear the accelerometer around their waist just above the right hip. Daily average minutes of moderate-to-vigorous physical activity, light physical activity, and sedentary behavior will be reported as a means of describing overall physical activity.
Epigenetic Profile | Baseline and After Study Week 12
  We will collect saliva and process this saliva according to established procedures for genomic DNA analyses--allowing for epigenetic profiling to occur.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary C Pope, PhD, Principal Investigator — University of Oklahoma Health Sciences; Mikhail Kellawan, PhD, Principal Investigator — University of Oklahoma, Department of Health and Exercise Science; Andriy Yabluchanskiy, MD, PhD, Principal Investigator — University of Oklahoma Health Sciences
Locations (1):
- University of Oklahoma Health Sciences, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pope ZC, Yabluchanskiy A, Mukli P, Robertson MC, Oliver JA, Borengasser SJ, Ratke MM, Matney JE, Mixon C, Henson C, Kellawan JM. Smartphone-Based Physical Activity Program to Reduce "Chemo-Brain" Symptoms and Improve Health in Cancer Survivors With and Without Type 2 Diabetes: Protocol for a Single-Arm Pre-Post Pilot Trial. JMIR Res Protoc. 2025 Dec 10;14:e79739. doi: 10.2196/79739. PMID 41370824